CLINICAL TRIAL: NCT02197754
Title: Adaptation in Polyphenol Bioavailability and Bioactivity During Long Term Exposure to Polyphenol-Rich Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS46
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: pharmacokinetics; polyphenol metabolites; lean individuals; obese individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polyphenol Diet (Experimental): After 2 weeks of adaptation to a controlled diet, polyphenol-rich fruits (berries and apple) and beverages (tea) will be fed (8 wks) as part of a controlled diet (10 wks total).
  Interventions: Other: Controlled diet

INTERVENTIONS:
Other: Controlled diet — Volunteers will be provided a controlled diet during the entirety of the 10 week treatment period. Meals will be prepared using traditional American foods.
  The controlled diet will include polyphenol-rich foods, including apples, berries, and green tea. A blend of multiple polyphenol-rich foods was chosen to investigate whole foods, multiple commodities, and multiple bioactives.

SUMMARY:
There are two primary objectives to be addressed in this study: to assess the differential response in bioavailability and metabolic pathways between lean and obese individuals exposed to acute, short term (14 day), and long-term (10-week) consumption of polyphenol-rich fruits (berries and apple), and beverages (tea); and to determine the differential systemic and gut anti-inflammatory response between obese and lean individuals exposed to polyphenol-rich fruits (berries and apple), and beverages (tea).

ELIGIBILITY:
Exclusion Criteria:

* Younger than 25 years old or older than 75 years old
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol (dicumarol), or Miradon (anisindione)
* Presence of any gastrointestinal disease, metabolic disease, bariatric surgery, or malabsorption syndromes that may interfere with the study goals
* Have been pregnant during the previous 12 months, are currently pregnant or lactating, or plan to become pregnant during the study
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides greater than 300 mg/dL
* Fasting glucose greater than 126 mg/dL
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months).
* Use of any tobacco products in past 3 months
* Unwillingness to abstain from herbal supplements for two weeks prior to the study and during the study
* Known (self-reported) allergy or adverse reaction to study foods
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Polyphenol metabolites - Wk 2 | 2 weeks after start of intervention
  Polyphenol metabolites will be measured in blood and urine after 2 weeks of a controlled diet.
Polyphenol metabolites - Wk 4 | 4 weeks after start of intervention
  Polyphenol metabolites will be measured in blood and urine after 4 weeks of a controlled diet. Weeks 3 and 4 will contain fruits and beverage rich in polyphenols.
Polyphenol metabolites - Wk 10 | 10 weeks after start of intervention
  Polyphenol metabolites will be measured in blood and urine after 10 weeks of a controlled diet. Weeks 3 through 10 will contain fruits and beverage rich in polyphenols.
Systemic inflammation - Wk 2 | 2 weeks after start of intervention
  Markers of inflammation (such as CRP, serum amyloid A, IL-6, IL-1B, TNF, and interferon-gamma will be measured.
Systemic Inflammation - Wk 4 | 4 weeks after start of intervention
  Markers of inflammation (such as CRP, serum amyloid A, IL-6, IL-1B, TNF, and interferon-gamma will be measured.
Systemic Inflammation - Wk 10 | 10 weeks after start of intervention
  Markers of inflammation (such as CRP, serum amyloid A, IL-6, IL-1B, TNF, and interferon-gamma will be measured.

SECONDARY OUTCOMES:
Gastrointestinal Health - Wk 2 | 2 weeks after start of intervention
  Gut permeability and inflammation will be measured in fecal samples.
Gastrointestinal Health - Wk 4 | Wk 4
  Gut permeability and inflammation will be measured in fecal samples.
Gastrointestinal Health - Wk 10 | 10 weeks after start of intervention
  Gut permeability and inflammation will be measured in fecal samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Beltsville Human Nutrition Center, Beltsville, Maryland, United States